CLINICAL TRIAL: NCT05844566
Title: Implementation of a Decision Support System and Its Effect on Early Optimisation of Lipid-Lowering Therapies in Patients With Acute Coronary Syndrome: a Cluster Randomised Controlled Trial
Brief Title: OptimiZation Of Lipid Lowering Therapies Using a Decision Support System In Patients With Acute Coronary Syndrome.
Acronym: ZODIAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Sanofi (Industry); Axtria, Inc. (Unknown); Hospital Universitario La Paz (Other); Hippocrates Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 22HH7982
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction
Keywords: Acute Coronary Syndrome; Decision Support System; Lipid Lowering Therapies; Low Density Lipoprotein; Heart Attack; ST Elevation Myocardial Infarction; Non-ST Elevation Myocardial Infarction; Coronary Disease
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Coronary Disease

STUDY DESIGN:
Intervention Model Description: Cluster randomised controlled trial. Study sites are randomised to intervention or no intervention.
Who Masked: Participant
Masking Description: The patient will be notified at the end of the study in regard to allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision Support System (DSS) (Other): Patients of this cohort are seen at a site randomised to the availability of the DSS. These patients will be provided routine clinical care including local/national prescribing guidelines during the course of the study. In addition to routine clinical care, the DSS which is available online, is a tool intended for clinicians to estimate the clinical benefit of any LLT regimen, whether monotherapy or combination therapies.
  Interventions: Device: Decision Support System (DSS)
- Non-Decision Support System (Non-DSS) (No Intervention): Patients of this cohort are seen at a site randomised to no availability of a DSS (Non-DSS). These patients will be provided routine clinical care including local / national prescribing guidelines during the course of the study.

INTERVENTIONS:
Device: Decision Support System (DSS) — This DSS will provide estimates of potential benefits in terms of ASCVD risk reduction (composite endpoint: combined non-fatal myocardial infarction, non-fatal ischaemic stroke and cardiovascular death) as a function of treatment duration and magnitude of LDL-C lowering.
  The DSS does not recommend treatments but shows the expected ASCVD risk, absolute and relative ASCDV risk reductions and number needed to treat for the various treatments selected by the clinical user on the potential value of initiation of an add-on therapy for reducing the risk of recurrent Cardiovascular (CV) events. Implementing the patient-specific recommendation remains at the clinicians' discretion.
  Arms: Decision Support System (DSS)

SUMMARY:
The goal of this clinical trial is to compare implementation of a Decision Support System (DSS) - aligned to the 2019 ESC/EAS Guidelines - in addition to routine clinical care versus routine clinical care without availability of a DSS, in participants aged ≥18 to < 80 years old presenting with Acute Coronary Syndrome (ACS).

The main questions it aims to answer are:

* to assess whether the availability of a DSS (which provides estimates of risk and estimates of potential benefit through LDL-C lowering) to current practice results in an increase in the early initiation of combination Lipid Lowering Therapies (LLTs) or intensification of LLT regimens compared to current practice alone over a 16-week period after an Acute Coronary Syndromes (ACS) event
* To estimate in the study cohort the potential benefits of guideline-based LLT intensification via simulation-based methods using estimates of baseline risk: LLT utilisation, additional LDL-C reductions and LDL-C goal achievement, on simulated risk of CV events through modelling.

Participants will give consent to randomised clinical sites to collect their data. The clinical sites will either be randomised to standard of care or the availability of and access to the DSS.

Researchers will compare patients from DSS and Non-DSS sites to see if the availability of the DSS results in implementation of more intensive lipid lowering regimens, resulting in the achievement of lower LDL-C values as well as the proportion of patients who reach target LDL-C levels (<1.4 mmol/L (<55 mg/dL) by Week 16.

DETAILED DESCRIPTION:
Patients with acute coronary syndromes (ACS) including myocardial infarction (MI) remain at risk of future cardiovascular events depending upon the interaction between inherited genetic factors/ and environmental factors including cholesterol over their lifetime. Expert guidelines on secondary prevention such as the ESC therefore increasingly recognise a more individualised approach.

Lowering LDL-C with high intensity lipid lowering therapies (LLTs) initiated within 10 days of an ACS reduces risk more than less intense regimens. In the SWEDEHEART registry which included 40,6007 patients over a median follow up of 3.78 years, patients who achieved the largest absolute reductions in LDL-C or greatest percentage reduction in LDL-C, had the lowest risk of a range of cardiovascular events and mortality. The approach to use of lipid lowering (LLT) was statin based monotherapy with few attaining the recommended cholesterol goals.

The 2019 European Society of Cardiology (ESC) and European Atherosclerosis Society (EAS) dyslipidaemia guidelines categorise patients with an ACS event as very-high risk and recommend an LDL-C goal of < 1.4 mmol/L (<55 mg/dL) and >50% reduction in LDL-C in this population. But several studies in European populations have highlighted gaps between clinical practice/ implementation of treatment recommendations compared with evidence based guideline recommendations. In the DA VINCI study representing 5,888 patients prescribed LLT in 18 European countries, LDL-C goal achievement in very-high risk populations was just 39% per 2016 ESC/EAS guidelines of<1.8mmol/L with only about 18% achieving the new recommended lower goal of <1.4mmol/L. It has become clear that greater implementation/ use of available combination therapies will be needed if lower recommended goals are to be achieved. It is unclear what the barriers are to earlier implementation and may include a lack of physician understanding of risk of further CV events or a lack of understanding of the quantifiable benefits from specific magnitudes of LDL-C lowering.

The aim of this trial is to assess whether providing information to those managing ACS patients that quantify absolute risk and the absolute benefit from different lipid lowering regimens through access to a Decision Support Tool (DSS) system is more likely to result in earlier intensification of lipid lowering regimens and thus result in a greater proportion of patients achieving the ESC lipid lowering goals after ACS compared to patients being managed routinely without access to a DSS standard (cluster RCT design). It is well established that unless treatments are initiated through secondary care or as part of acute care pathways, there is considerable inertia in further optimisation of treatment in primary care. Thus, this trial will assess whether presenting quantifiable data on risks and benefits results in behaviour change among secondary care physicians and improves cholesterol management within 4 months of an ACS.

The DSS is available online or remotely accessible via a website intended for clinicians to estimate the clinical benefit of any LLT regimen, whether single or combination therapies. The DSS shows the expected risk, risk reductions and number needed to treat for the various treatments selected by the clinical user on the potential value of initiation of an add-on therapy for reducing the risk of other Cardiovascular (CV) events. This DSS provides a graphical and tabular representation of the time-dependent CV treatment benefit model for LLTs published in a peer-reviewed journal article.

The trial hypothesises that having a pictorial representation of both individual risk and recommended treatments will encourage clinicians to implement clinical guidelines more closely. The clinicians using the DSS will be asked to complete a DSS evaluation at the end of the trial. Implementing the patient-specific recommendation remains at the clinicians' discretion.

ELIGIBILITY:
Inclusion criteria:

Sites:

* Manage ACS patients as defined by: Symptoms of myocardial ischemia with an unstable pattern, occurring at rest or with minimal exertion, within 72 hours of an unscheduled hospital admission due to presumed or proven obstructive coronary disease and at least one of the following:

  * Elevated cardiac biomarkers
  * Resting electrocardiographic changes consistent with ischemia or infarction, plus additional evidence of obstructive coronary disease from regional wall motion or perfusion abnormality, 70% or more epicardial coronary stenosis by angiography, or need for coronary revascularization procedure
* Mange post ACS follow up care of patients including risk factor control
* Ability to provide follow up information on patient care for a minimum of 16 weeks including blood tests
* Willing/ able to access and undertake training for the DSS
* Adequate internet connection at site and the ability to access the DSS
* No restrictions on use of LLTs (within national guidelines/ reimbursement)
* Ability to include all essential parameters and patient information for DSS input

Participants:

* Aged ≥18 to < 80 years old
* Provide written informed consent
* Presenting to a study site with ACS as LLT naïve, monotherapy or combination therapy (defined as more than one LLT agent)
* Willing to take lipid lowering treatments for the secondary prevention of cardiovascular disease
* Attending the same study site (or same clinical team) for ACS follow up to ensure follow up data can be collected; or ensure that follow up data can be collected from other clinical institutions as part of the clinical pathway.

Exclusion criteria:

Sites:

* Unable to capture/ provide data on patients with ACS during admission and follow up
* Unable or unwilling to use lipid lowering treatments other than statins for ACS care

Participants:

* Unable to provide written informed consent
* LDL-C measurement < 1.8 mmol/L at admission

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1139 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Optimisation of the intensity of Lipid Lowering Therapy within 16 weeks of index ACS | 16 weeks
  Proportion of patients treated with combination therapy, or who receive escalated monotherapy, or escalated combination therapy, within 16 weeks of the index ACS.

SECONDARY OUTCOMES:
Time to initiation | 16 weeks
  Time to initiation of combination therapy or escalation of Lipid lowering therapy as defined in the primary endpoint
LDL-C Level | 16 weeks
  LDL-C by Week 16
Target LDL-C reduction | 16 weeks
  Proportion of patients reaching target LDL-C level (<1.4 mmol/L (<55 mg/dL) by Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Kausik Ray, Professor, Principal Investigator — Imperial College London
Locations (42):
- Italy (11):
  - AUSL di Bologna-Ospedale Maggiore, Bologna
  - Azienda Ospedaliera di Rilievo Nazionale (A.O.R.N.) "Sant'Anna e San Sebastiano" di Caserta, Caserta
  - A.O.U. Ospedali Riuniti U.O.C. Cardiologia e UTIC, Foggia
  - IRCCS. A.O.U. Policlinico San Martino IST, Genova
  - Azienda Ospedaliera Universitaria Gaetano Martino, Messina
  - IRCCS Policlinico San Donato, Milan
  - A.O.U Policlinico di Modena S.C. di Cardiologia, Modena
  - Ospedale di Cisanello - A.U.O.P. Azienda Ospedaliera Universitaria, Pisa
  - AUSL-IRCCS di Reggio Emilia, Reggio Emilia
  - Ospedale Sandro Pertini - ASL Roma 2, Roma
  - Azienda Ospedaliero Universitaria Santa Maria della Misericordia, Udine
- Spain (14):
  - Hospital Clínico Universitario Santiago de Compostela, Santiago de Compostela, A Coruña
  - University Hospital of A Coruña, A Coruña, Coruña
  - Hospital HM Montepríncipe, Boadilla del Monte, Madrid
  - Puerta de Hierro Majadahonda University Hospital, Majadahona, Madrid
  - Hospital Universitario Rey Juan Carlos, Móstoles, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario La Luz Quiron, Madrid
  - Gregorio Marañón General University Hospital, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen Macarena, Seville
- United Kingdom (17):
  - Luton and Dunstable University Hospital, Luton, Bedfordshire
  - Glan Glwyd Hospital, Bodelwyddan, Denbighshire
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - Conquest Hospital, Brighton, East Sussex
  - Scunthorpe General Hospital, Scunthorpe, North Lincolnshire
  - Kettering General Hospital, Kettering, Northamptonshire
  - Southern Health and Social Care Trust, Craigavon Area Hospital, Portadown, Northen Ireland
  - Royal United Hospital, Bath, Somerset
  - Freeman Hospital, Newcastle upon Tyne, Tyne and Wear
  - North Tyneside General Hospital, North Shields, Tyne and Wear
  - Sunderland Royal Hospital, Sunderland, Tyne and Wear
  - Sandwell General Hospital, Birmingham, West Midlands
  - Russell's Hall Hospital, Dudley, West Midlands
  - Worthing Hospital, Worthing, West Sussex
  - Calderdale Royal Hospital, Halifax, West Yorkshire
  - Worcestershire Royal Hospital, Worcester, Worcestershire
  - Hammersmith Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schubert J, Lindahl B, Melhus H, Renlund H, Leosdottir M, Yari A, Ueda P, James S, Reading SR, Dluzniewski PJ, Hamer AW, Jernberg T, Hagstrom E. Low-density lipoprotein cholesterol reduction and statin intensity in myocardial infarction patients and major adverse outcomes: a Swedish nationwide cohort study. Eur Heart J. 2021 Jan 20;42(3):243-252. doi: 10.1093/eurheartj/ehaa1011. PMID 33367526
- [Background] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; ESC Scientific Document Group. 2018 ESC/ESH Guidelines for the management of arterial hypertension. Eur Heart J. 2018 Sep 1;39(33):3021-3104. doi: 10.1093/eurheartj/ehy339. No abstract available. PMID 30165516
- [Background] Mach F, Baigent C, Catapano AL, Koskinas KC, Casula M, Badimon L, Chapman MJ, De Backer GG, Delgado V, Ference BA, Graham IM, Halliday A, Landmesser U, Mihaylova B, Pedersen TR, Riccardi G, Richter DJ, Sabatine MS, Taskinen MR, Tokgozoglu L, Wiklund O; ESC Scientific Document Group. 2019 ESC/EAS Guidelines for the management of dyslipidaemias: lipid modification to reduce cardiovascular risk. Eur Heart J. 2020 Jan 1;41(1):111-188. doi: 10.1093/eurheartj/ehz455. No abstract available. PMID 31504418
- [Background] Bohula EA, Morrow DA, Giugliano RP, Blazing MA, He P, Park JG, Murphy SA, White JA, Kesaniemi YA, Pedersen TR, Brady AJ, Mitchel Y, Cannon CP, Braunwald E. Atherothrombotic Risk Stratification and Ezetimibe for Secondary Prevention. J Am Coll Cardiol. 2017 Feb 28;69(8):911-921. doi: 10.1016/j.jacc.2016.11.070. PMID 28231942
- [Background] Ference BA, Ginsberg HN, Graham I, Ray KK, Packard CJ, Bruckert E, Hegele RA, Krauss RM, Raal FJ, Schunkert H, Watts GF, Boren J, Fazio S, Horton JD, Masana L, Nicholls SJ, Nordestgaard BG, van de Sluis B, Taskinen MR, Tokgozoglu L, Landmesser U, Laufs U, Wiklund O, Stock JK, Chapman MJ, Catapano AL. Low-density lipoproteins cause atherosclerotic cardiovascular disease. 1. Evidence from genetic, epidemiologic, and clinical studies. A consensus statement from the European Atherosclerosis Society Consensus Panel. Eur Heart J. 2017 Aug 21;38(32):2459-2472. doi: 10.1093/eurheartj/ehx144. PMID 28444290
- [Background] Khan I, Peterson ED, Cannon CP, Sedita LE, Edelberg JM, Ray KK. Time-Dependent Cardiovascular Treatment Benefit Model for Lipid-Lowering Therapies. J Am Heart Assoc. 2020 Aug 4;9(15):e016506. doi: 10.1161/JAHA.120.016506. Epub 2020 Jul 28. PMID 32720582
- [Background] Ray KK, Reeskamp LF, Laufs U, Banach M, Mach F, Tokgozoglu LS, Connolly DL, Gerrits AJ, Stroes ESG, Masana L, Kastelein JJP. Combination lipid-lowering therapy as first-line strategy in very high-risk patients. Eur Heart J. 2022 Feb 22;43(8):830-833. doi: 10.1093/eurheartj/ehab718. No abstract available. PMID 34636884
- [Background] Ray KK, Molemans B, Schoonen WM, Giovas P, Bray S, Kiru G, Murphy J, Banach M, De Servi S, Gaita D, Gouni-Berthold I, Hovingh GK, Jozwiak JJ, Jukema JW, Kiss RG, Kownator S, Iversen HK, Maher V, Masana L, Parkhomenko A, Peeters A, Clifford P, Raslova K, Siostrzonek P, Romeo S, Tousoulis D, Vlachopoulos C, Vrablik M, Catapano AL, Poulter NR; DA VINCI study. EU-Wide Cross-Sectional Observational Study of Lipid-Modifying Therapy Use in Secondary and Primary Care: the DA VINCI study. Eur J Prev Cardiol. 2021 Sep 20;28(11):1279-1289. doi: 10.1093/eurjpc/zwaa047. PMID 33580789
- [Background] Steen DL, Khan I, Ansell D, Sanchez RJ, Ray KK. Retrospective examination of lipid-lowering treatment patterns in a real-world high-risk cohort in the UK in 2014: comparison with the National Institute for Health and Care Excellence (NICE) 2014 lipid modification guidelines. BMJ Open. 2017 Feb 17;7(2):e013255. doi: 10.1136/bmjopen-2016-013255. PMID 28213597
- [Background] Ferrieres J, Gorcyca K, Iorga SR, Ansell D, Steen DL. Lipid-lowering Therapy and Goal Achievement in High-risk Patients From French General Practice. Clin Ther. 2018 Sep;40(9):1484-1495.e22. doi: 10.1016/j.clinthera.2018.07.008. Epub 2018 Aug 18. PMID 30126705
- [Background] Arca M, Ansell D, Averna M, Fanelli F, Gorcyca K, Iorga SR, Maggioni AP, Paizis G, Tomic R, Catapano AL. Statin utilization and lipid goal attainment in high or very-high cardiovascular risk patients: Insights from Italian general practice. Atherosclerosis. 2018 Apr;271:120-127. doi: 10.1016/j.atherosclerosis.2018.02.024. Epub 2018 Feb 17. PMID 29499359
- [Background] Blaum C, Seiffert M, Gossling A, Kroger F, Bay B, Lorenz T, Braetz J, Graef A, Zeller T, Schnabel R, Clemmensen P, Westermann D, Blankenberg S, Brunner FJ, Waldeyer C. The need for PCSK9 inhibitors and associated treatment costs according to the 2019 ESC dyslipidaemia guidelines vs. the risk-based allocation algorithm of the 2017 ESC consensus statement: a simulation study in a contemporary CAD cohort. Eur J Prev Cardiol. 2021 Mar 23;28(1):47-56. doi: 10.1093/eurjpc/zwaa088. PMID 33580772
- [Background] Marz W, Dippel FW, Theobald K, Gorcyca K, Iorga SR, Ansell D. Utilization of lipid-modifying therapy and low-density lipoprotein cholesterol goal attainment in patients at high and very-high cardiovascular risk: Real-world evidence from Germany. Atherosclerosis. 2018 Jan;268:99-107. doi: 10.1016/j.atherosclerosis.2017.11.020. Epub 2017 Nov 20. PMID 29197254
- [Background] Kuiper JG, Sanchez RJ, Houben E, Heintjes EM, Penning-van Beest FJA, Khan I, van Riemsdijk M, Herings RMC. Use of Lipid-modifying Therapy and LDL-C Goal Attainment in a High-Cardiovascular-Risk Population in the Netherlands. Clin Ther. 2017 Apr;39(4):819-827.e1. doi: 10.1016/j.clinthera.2017.03.001. Epub 2017 Mar 27. PMID 28347514
- [Background] Koskinas KC, Gencer B, Nanchen D, Branca M, Carballo D, Klingenberg R, Blum MR, Carballo S, Muller O, Matter CM, Luscher TF, Rodondi N, Heg D, Wilhelm M, Raber L, Mach F, Windecker S. Eligibility for PCSK9 inhibitors based on the 2019 ESC/EAS and 2018 ACC/AHA guidelines. Eur J Prev Cardiol. 2021 Mar 23;28(1):59-65. doi: 10.1177/2047487320940102. Epub 2020 Jul 20. PMID 33755142
- [Background] Allahyari A, Jernberg T, Hagstrom E, Leosdottir M, Lundman P, Ueda P. Application of the 2019 ESC/EAS dyslipidaemia guidelines to nationwide data of patients with a recent myocardial infarction: a simulation study. Eur Heart J. 2020 Oct 21;41(40):3900-3909. doi: 10.1093/eurheartj/ehaa034. PMID 32072178
- [Background] Mancia G, Rea F, Corrao G, Grassi G. Two-Drug Combinations as First-Step Antihypertensive Treatment. Circ Res. 2019 Mar 29;124(7):1113-1123. doi: 10.1161/CIRCRESAHA.118.313294. PMID 30920930
- [Background] Dorresteijn JA, Visseren FL, Wassink AM, Gondrie MJ, Steyerberg EW, Ridker PM, Cook NR, van der Graaf Y; SMART Study Group. Development and validation of a prediction rule for recurrent vascular events based on a cohort study of patients with arterial disease: the SMART risk score. Heart. 2013 Jun;99(12):866-72. doi: 10.1136/heartjnl-2013-303640. Epub 2013 Apr 10. PMID 23574971
- [Background] McKay AJ, Gunn LH, Ference BA, Dorresteijn JAN, Berkelmans GFN, Visseren FLJ, Ray KK. Is the SMART risk prediction model ready for real-world implementation? A validation study in a routine care setting of approximately 380 000 individuals. Eur J Prev Cardiol. 2022 Mar 30;29(4):654-663. doi: 10.1093/eurjpc/zwab093. PMID 34160035
- [Background] Gao F, Earnest A, Matchar DB, Campbell MJ, Machin D. Sample size calculations for the design of cluster randomized trials: A summary of methodology. Contemp Clin Trials. 2015 May;42:41-50. doi: 10.1016/j.cct.2015.02.011. Epub 2015 Mar 9. PMID 25766887
- [Background] Campbell MK, Piaggio G, Elbourne DR, Altman DG; CONSORT Group. Consort 2010 statement: extension to cluster randomised trials. BMJ. 2012 Sep 4;345:e5661. doi: 10.1136/bmj.e5661. No abstract available. PMID 22951546
- [Background] Bellamy SL, Gibberd R, Hancock L, Howley P, Kennedy B, Klar N, Lipsitz S, Ryan L. Analysis of dichotomous outcome data for community intervention studies. Stat Methods Med Res. 2000 Apr;9(2):135-59. doi: 10.1177/096228020000900205. PMID 10946431
- [Background] Campbell MJ, Donner A, Klar N. Developments in cluster randomized trials and Statistics in Medicine. Stat Med. 2007 Jan 15;26(1):2-19. doi: 10.1002/sim.2731. PMID 17136746
- [Background] Parker RA, Weir CJ. Multiple secondary outcome analyses: precise interpretation is important. Trials. 2022 Jan 10;23(1):27. doi: 10.1186/s13063-021-05975-2. PMID 35012627
- [Background] Cannon CP, Khan I, Klimchak AC, Reynolds MR, Sanchez RJ, Sasiela WJ. Simulation of Lipid-Lowering Therapy Intensification in a Population With Atherosclerotic Cardiovascular Disease. JAMA Cardiol. 2017 Sep 1;2(9):959-966. doi: 10.1001/jamacardio.2017.2289. PMID 28768335
- [Background] Rubin, M. When to adjust alpha during multiple testing: a consideration of disjunction, conjunction, and individual testing. Synthese 199, 10969-11000 (2021).
- [Background] Ritz J, Spiegelman D. Equivalence of conditional and marginal regression models for clustered and longitudinal data. Statistical Methods in Medical Research. 2004;13(4):309-323. doi:10.1191/0962280204sm368ra
- See also: Framework to aid in the creation of apps across multiple platforms including iOS, Android and Windows. — http://cordova.apache.org/
- See also: Angular is a development platform, built on TypeScript. This link can help you understand Angular: what Angular is, what advantages it provides, and what you might expect as you start to build applications — http://angular.io/guide/what-is-angular
- See also: Empirical estimates of ICCs from changing professional practice studies. (Very small ICCs rounded to 0.0001; Negative ICCs truncated at zero; n/a = not applicable). — https://www.abdn.ac.uk/hsru/documents/iccs-web.xls